CLINICAL TRIAL: NCT04733898
Title: Social Health Games: a Gamified Intervention to Decrease Loneliness in Older Adults - a Randomized Controlled Trial
Brief Title: Social Health Games: The Use of Online Games to Decrease Loneliness in Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Aimed sample size could not be reached within the time that was taken for recruitment.
Sponsor: Radboud University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-6884; 645.003.002 (Other Grant/Funding Number: NWO)
Record Dates: First submitted 2021-01-28; First posted 2021-02-02 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2021-01

CONDITIONS: Loneliness
Keywords: Social network; Digital technology; Social games

STUDY DESIGN:
Intervention Model Description: Three different groups will start simultaneously, with each participant in one and only one condition.
Who Masked: Investigator
Masking Description: The investigator analyzing data will be blind to the group coding and the personal information. Only anonymized data will be available to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social games (Experimental): Participants in the social games group will be given access to an app with games that are either adaptations of well-known games or newly developed games, all designed to be played with just text messages and photos. A game is essentially a chat group with the people you invited to play that specific game with. Participants can play with their own network of family and friends, as well as other people in the same condition.
  Interventions: Other: SamenSpelen.app
- Non-personal games (Active Comparator): Participants in the active control group will be given access to an app that offers 'non-personal games'. The portal will contain a subset of the social games, which have been adapted for non-personal play. This means that all aspects that make the games personal are removed and discouraged. The games that remain can still be played with others (family/friends and others in the same condition), but are designed not to elicit personal interaction. Participants are asked to play the games at least twice a week, but may play as often as they like.
  Interventions: Other: FijnSpelen.app
- Passive control (No Intervention): The passive control group will be given access to an app that contains no games. Similar to the other groups, the portal is used to complete the questionnaires. Use of other games, (gaming) apps or social media platforms is allowed in this group, as in the other groups. The only restriction they will not have access to the games offered in the social games and active control groups.

INTERVENTIONS:
Other: SamenSpelen.app — An app designed to play simple, social games in a chat environment. These games are designed to elicit personal interaction.
  Arms: Social games
Other: FijnSpelen.app — An app designed to play simple, social games in a chat environment. These games are designed to not elicit personal interaction.
  Arms: Non-personal games

SUMMARY:
This study examines whether social platform games are effective in expanding the social network and decreasing the experienced levels of loneliness in older adults. The newly developed social games will be compared to non-personal games and not playing games.

DETAILED DESCRIPTION:
Rationale: loneliness and social isolation are an increasing problem in older adults with the aging of society. One option to foster social contact is through online games, which allow social interaction at a distance.

Objective: to investigate whether playing social online games has a beneficial effect on subjective loneliness and social network in older adults, compared with playing non-personal games and not playing games.

Study design: 3-arm randomized controlled trial.

Study population: A sample of 300 human volunteers aged 65 and over, who have access to a smartphone and an internet connection. The sample will be evenly distributed across the three groups.

Everybody else is allowed to use the gaming portal; they will form the pool of people that the participants can play with. This pool will be tracked within the gaming portal and posed some questions regarding their fellow players and their experiences loneliness. People aged under 16 can play but will not be tracked.

Intervention (if applicable): Three groups: (I) Intervention group, who will be given access to an app with the social games, and are encouraged to use this app as much as possible, (II) active control group, who will be given access to an app with non-personal games, and are encouraged to use this app as much as possible, (III) passive control group, who will be given access to an app with no games. The platform has a chatbot designed to take the questionnaires.

Comparison between groups (I+II) and (III) will show whether playing games has an effect on loneliness/social network.

Comparison between groups (I) and (II) will show whether the social aspect of games has additional benefits over solo-games on loneliness/social network.

Main study parameters/endpoints: Primary outcome: change in perceived loneliness over time; secondary outcomes: change in (I) social network composition and (II) health-related outcomes over time. All acquired via chatbot questionnaires.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: the participants will have to download and install the app. Participants in the social games group will be invited to play games with people from their own network and may plan as often as they want with whom they want, but are encouraged to play at least twice a week. Participants in the non-personal games group will be invited to play games as often as they want but are encouraged to play at least twice a week. All participants are asked to complete questionnaires. In-app questionnaires will be administered monthly: the complete set of questionnaires at baseline, after 6 months, and after 12 months (duration 1.5 hours), and the loneliness questionnaire monthly (duration 10 minutes) Since the questionnaires contain questions on loneliness and mental wellbeing, some might be perceived as sensitive.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* Have access to a smartphone with an internet connection

Exclusion Criteria:

* Visual or cognitive impairments that limit independent use of a mobile phone
* Not being fluent in the Dutch language

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Loneliness indirect | Three months
  The change in indirectly measured loneliness (De Jong Gierveld loneliness scale (range 1-11, higher indicating more loneliness)) over three months between the three groups
Loneliness direct | Three months
  The change in directly measured loneliness (Likert scale (range 1-5, higher indicating more loneliness) over three months between the three groups

SECONDARY OUTCOMES:
Loneliness time series | Twelve months
  The temporal variability in indirectly measured loneliness (De Jong Gierveld loneliness scale (range 1-11, higher indicating more loneliness)) over twelve months
Wellbeing | Twelve months
  The change in wellbeing (SPF-IL) between the groups over twelve months
Social network composition | Twelve months
  The change in social network composition (NESTOR-LSN) between the groups over twelve months

OTHER OUTCOMES:
Gaming behaviour and social interactions | Twelve months
  Data on the games participants play (retrieved from the backend game data), when and with whom they play them (retrieved from questionnaires assessed after games have been played. Questions on relationship type and intensity have been adapted from the NESTOR-LSN questionnaire.)

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Olde Rikkert, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anonymized questionnaire and backend game data will be stored in the repisitory of the Data Archiving and Networked Services (DANS-Easy) after finalizing the project and all data analyses. After that, it is available open access.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the end of the project (Mid 2024).
Access Criteria: Open Access

REFERENCES:
- See also: The project website (in Dutch), including information on the study — http://www.samenspelen.online